CLINICAL TRIAL: NCT07019077
Title: Incidence of Late Haemorrhage After Invasive Gastroenterological Endoscopic Manoeuvre in Patients Treated With Anticoagulants Compared to Non-anticoagulated Patients
Acronym: EMOSCOPIO
Status: Recruiting | Type: Observational
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Humanitas Research Hospital IRCCS, Rozzano-Milan (Other); Valduce Hospital (Other); Azienda Ospedaliera di Lecco (Other); Istituto Auxologico Italiano (Other); Università degli Studi dell'Insubria (Other); ASST Sette Laghi (Other)
Responsible Party: Principal Investigator, Barbara Scimeca, Principal Investigator - Medical Doctor, Centro Cardiologico Monzino
Other Study IDs: L2-223
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Bleeding
Keywords: endoscopic gastroenterological manoeuvre
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients on oral anticoagulant therapy with vitamin K antagonists (AVKs; warfarin and acenocoumarol) and direct oral anticoagulants (DOACs; apixaban, dabigatran, edoxaban and rivaroxaban), are advised to consider discontinuing treatment in anticipation of invasive manoeuvres. Guidelines and expert consensus recommend, in clinical conditions with a high risk of bleeding, to suspend oral anticoagulant treatment with DOACs 2 or 3 days before the procedure, depending on the glomerular filtrate, to suspend warfarin from day -5 and acenocoumarol from day -4, and to introduce heparins from day -3 after discontinuation of AVKs (so-called 'bridging therapy') for manoeuvres with a high risk of bleeding. In manoeuvres with a low bleeding risk it is possible not to suspend the anticoagulant or to reduce its intensity. Obviously, the patient's intrinsic haemorrhagic and thrombotic risk (antiplatelet intake, renal insufficiency, hepatopathy, age, mechanical valve prosthesis, oncological condition, etc.) must also be taken into account in the overall assessment of pre-procedural preparation.

Gastroenterological endoscopic manoeuvres are generally considered to be at low haemorrhagic risk even if biopsy is planned, but are at high haemorrhagic risk if polypectomy or mucosectomy is planned. The most complex problem arises at the time of re-introduction of anticoagulant post-procedure. In fact, studies evaluating this specific aspect are very few and heterogeneous and mostly retrospective. The variables that are associated with an increased risk of bleeding are: the number and site of polypectomies, the diameter of the polyps, and local haemostasis techniques. Late haemorrhages (>24 hours) are of concern because the patient is generally at home and because, by the time the eschar falls out (varying between 4 and 10 days post-procedure), they have already resumed anticoagulation. However, there are no prospective studies of sufficient number to clarify whether the reintroduction of anticoagulation modifies the haemorrhagic risk, when is the time of greatest risk after the procedure, and which variables associated with the patient and the procedure most modify the haemorrhagic risk.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Expected endoscopic manoeuvre among those listed below
* EGDS ± biopsy/polypectomy
* Colonoscopy ± biopsy/polypectomy
* Echoguided endoscopy ± biopsy/polypectomy
* Double-balloon enteroscopy
* ERCP (endoscopic retrograde cholangio-pancreatography) ± sphincterotomy

Exclusion Criteria:

* Age < 18 years
* Known active neoplasms of the gastroenteric tract
* Gastrointestinal procedures performed as an emergency
* Patients with an intrinsic haemorrhagic diathesis (e.g. known plateletopenia < 50,000/mmc)
* Patients on antiplatelet treatment with clopidogrel or other thienopyridines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with/without anticoagulant treatment who are candidates for gastroenterological endoscopic procedures, either at low haemorrhagic risk (<1%) or at high haemorrhagic risk (>=1%).
Sampling Method: Non-Probability Sample
Enrollment: 4719 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of late bleeding | 30 days after the manoeuvre.
  The primary objective is to assess the incidence of late (>24 hours) bleeding from the gastro-enteric tract in anticoagulated patients after low and high risk endoscopic manoeuvres and to compare it with that observed in non-anticoagulated patients in the first 30 days after the manoeuvre.

SECONDARY OUTCOMES:
Incidence of early bleeding | First 24 hours
  Secondary objectives:
  * Incidence of early bleeding (first 24 hours) in relation to pre-procedural withdrawal or no withdrawal
  * Possible difference in bleeding incidence by anticoagulant class (AVK vs DOAC vs heparin)
  * Possible difference in bleeding incidence by type of endoscopic manoeuvre (low or high risk of bleeding)
  * Possible difference in bleeding incidence by mode of reintroduction of anticoagulant therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Cardiologico Monzino; IRCCS, Milan, Italy